CLINICAL TRIAL: NCT00152685
Title: High Dose Hyperoncotic Serum Albumin for the Treatment of the Acute Phase of Severe Head Injury
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: CP 02-04
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-09

CONDITIONS: Severe Head Injury
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Serum Albumin, Human

INTERVENTIONS:
Drug: human serum albumin

SUMMARY:
Experimentally high dose of hyperoncotic human serum albumin improve neurological recovery after head injury reduce cerebral edema and normalize apparent diffusion coefficient of water after ischemia reperfusion. The main hypothesis is that early administration of hyperoncotic serum albumin is able to reduce intracranial pressure for several days after severe head injury and thus reduce mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* severe head injury (GCS < 9) Next of kin informed consent

Exclusion Criteria:

* Cranio cerebral wound Pregnancy Hypoxemia (PaO2/FiO2< 300 mmHg) Blood loss > 1/2 blood mass Renal or cardiac failure,uncontrolled hypertension Head injury dating from more than 24 hours at the time of inclusion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40

PRIMARY OUTCOMES:
Reduction of the daily median value of intracranial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ter Minassian Aram, MD, PhD, Principal Investigator — Universitary hospital of Angers; Audibert Gérard, MD, PhD, Study Chair — Universitary hospital of Nancy; Vigue Bernard, MD, PhD, Study Chair — Universitary hospital of Le Kremlin Bicêtre
Locations (3):
- France (3):
  - Surgical intensive care. CHU, Angers, Cedex 9
  - Neurosurgical intensive care. CHU Le Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Neurosurgical intensive care. CHU de Nancy, Nancy